CLINICAL TRIAL: NCT06475469
Title: Description of the Immune Deficiency in Patients With Untreated Chronic Lymphocytic Leukemia and Search for Predictive Factors of Infectious Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PO22063
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Immunodeficiency; Lymphocyte subpopulations; Bronchiectasis
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Immunologic Deficiency Syndromes; Bronchiectasis | interventions — Blood Specimen Collection; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with untreated Chronic Lymphocytic Leukemia (CLL) (Other)
  Interventions: Biological: Blood sampling & Chest CT without injection

INTERVENTIONS:
Biological: Blood sampling & Chest CT without injection — Anlaysis of the repartition of non-tumorous lymphocytic subpopulation in patients with untreated Chronic Lymphocytic Leukemia (CLL)

SUMMARY:
Chronic Lymphocytic Leukemia (CLL) is the most common adult leukemia in western countries. CLL is most often discovered incidentally when a blood test carried out for another reason highlights an increase of subpopulation of white cells called lymphocytes. It is also sometimes diagnosed when complications such as an increase in the size of the lymph nodes or a decrease in other blood lines (red blood cells and platelets) occur. Its evolution is heterogeneous and only patients with symptoms require treated. CLL is aso characterized by its hability to induce immunodeficiency, which tends to worsen over time, even in patients who do not receive any treatment. Thus, patients with CLL have more infections than the general population, and these infectious complications are the leading cause of death. Similarly, vaccination, whether directed against classical pathogens such as influenzae or more recently against SARS-CoV2, is less effective in patients with CLL. The causes of this immune deficiency are not completely elucidated and the objective of our study is to analyze different subpopulations of lymphocytes thanks to a blood sample. The investigators thus hope to be able to determine more precisely the reasons underlying these infections in order to better prevent them.

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL) is a monoclonal B-cell proliferation and the most common leukemia of adults. It is characterized by infiltration of the bone marrow, lymph nodes and blood by small mature lymphocytes. It is an incurable pathology but its evolution is extremely heterogeneous. Thus, some patients will have a life expectancy close to normal without treatment, while for others, a progression of the disease will require the introduction of a specific treatment.

One of the main characteristics of CLL is the associated immune dysfunction. The presence of an increased risk of infectious complications has been clearly demonstrated, even in patients with indolent forms of the disease. Immunosuppression is multifactorial, affecting both humoral and cellular immunity. Nevertheless, the major abnormality associated with infectious risk in CLL is hypogammaglobulinemia. Hypogammaglobulinemia is present in approximately 20% of patients at diagnosis and worsens during the course of the disease. In particular, it is responsible for an impaired vaccine response and the occurrence of encapsulated bacterial infections. As with primary humoral immunodeficiency, chronic humoral immunodeficiency secondary to CLL is associated with the development of irreversible bronchiectasis, the prevalence of which is not well understood, and which increases the risk of severe respiratory infectious complications.

In CLL patients, the normal B lymphocyte compartment and in particular certain populations of interest such as the memory B lymphocyte populations have only been studied to a limited extent. Similarly, there is little data on follicular helper T cells (TfH cells) which play a key role in the acquisition of anti-infectious and particularly post-vaccination immunity.

The primary objective of this study is to analyze the distribution of non-tumor lymphocyte subpopulations in patients with untreated CLL

The secondary objectives of the research are:

1. To prospectively assess the frequency and severity of infections in patients with CLL
2. To search for an association between biological and particularly immunophenotypic data and the occurrence of infections
3. To define the prevalence of bronchiectasis in CLL patients
4. To study the clinical, immunological and biochemical factors associated with the presence of bronchiectasis in CLL patients

75 untreated CLL patients will be included in this study. Thoracic CT scan and immunophenotyping will be performed at inclusion. Infectious complications will be collected prospectively through a follow-up booklet provided to the patient at the time of inclusion. All infections requiring at least one consultation with the general practitioner will be collected. Reported infections will be graded according to a classification derived from the CTCAE.

Our study should help to better characterize the immune deficiency associated with CLL through the analysis of lymphocyte subpopulations. A better understanding of the mechanisms underlying this immune deficiency could lead to a better identification of patients at risk of infectious complications and to a better understanding of the vaccine efficacy deficit in CLL patients. Finally, earlier diagnosis and identification of patient profiles more likely to have bronchiectasis could allow for targeted and personalized therapeutic management and follow-up for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Untreated CLL patients
* Patients > 18 years of age
* Patients agreing to participate to the study
* Patients inured under the french social security system

Exclusion Criteria:

* Previously treated CLL patients
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Immunophenotyping | At inclusion
  Description of some circulating B and T cell subsets

SECONDARY OUTCOMES:
Bronchectasies | At inclusion
  presence of bronchiectasis (Non-contrast thin section thoracic CT-scan allowing to detect the ) and if present the severity index (Bhalla score)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France